CLINICAL TRIAL: NCT03475290
Title: Efficacy of Internet-Based Intervention for Occupational Stress Among Medical Professionals: A Randomized Controlled Trial
Brief Title: Internet-Based Intervention for Occupational Stress Among Medical Professionals
Acronym: Med-Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: Linkoeping University (Other Government); Stockholm University (Other)
Responsible Party: Principal Investigator, Ewelina Smoktunowicz, Principal Investigator, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I.N.16 Med-Stress
Record Dates: First submitted 2018-02-28; First posted 2018-03-23 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Stress, Psychological, Occupational; Burnout, Professional
Keywords: e-mental health; stress; burnout; self-efficacy; social support
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-Efficacy and Perceived Social Support (Experimental)
  Interventions: Behavioral: Personal resources' enhancement: self-efficacy and perceived social support
- Perceived Social Support and Self-Efficacy (Experimental)
  Interventions: Behavioral: Personal resources' enhancement: perceived social support and self-efficacy
- Self-Efficacy (Active Comparator)
  Interventions: Behavioral: Personal resources' enhancement: self-efficacy
- Perceived Social Support (Active Comparator)
  Interventions: Behavioral: Personal resources' enhancement: perceived social support

INTERVENTIONS:
Behavioral: Personal resources' enhancement: self-efficacy and perceived social support — The condition reflects cultivation hypothesis and consists of 2 sequential modules with self-efficacy enhancement module (SE) preceding perceived social support enhancement module (SS). Each module is comprised of 3 evidence-based, CBT-framed exercises: 1) SE: mastery experience, vicarious experience, and action planning, 2) SS: received support & cognitive distortions, social skills & peer support, action planning. Participants will have an option to engage in one or more out of four additional modules: relaxation, cognitive reconstruction, mindfulness, and lifestyle. The condition takes 6 weeks, 1 week per exercise.
  Arms: Self-Efficacy and Perceived Social Support
Behavioral: Personal resources' enhancement: perceived social support and self-efficacy — The condition reflects enabling hypothesis and consists of 2 sequential modules with perceived social support enhancement module (SS) preceding self-efficacy enhancement module (SE). Each module is comprised of 3 evidence-based, CBT-framed exercises: 1) SS: received support & cognitive distortions, social skills & peer support, and action planning, 2) SE: mastery experience, vicarious experience, and action planning. Participants will have an option to engage in one or more out of four additional modules: relaxation, cognitive reconstruction, mindfulness, and lifestyle. The condition takes 6 weeks, 1 week per exercise.
  Arms: Perceived Social Support and Self-Efficacy
Behavioral: Personal resources' enhancement: self-efficacy — The condition consists of self-efficacy enhancement module (SE) and is comprised of 3 evidence-based, CBT-framed exercises: mastery experience, vicarious experience, and action planning. Participants will have an option to engage in one or more out of four additional modules: relaxation, cognitive reconstruction, mindfulness, and lifestyle. The condition takes 3 weeks, 1 week per exercise.
  Arms: Self-Efficacy
Behavioral: Personal resources' enhancement: perceived social support — The condition consists of perceived social support enhancement module (SS) and is comprised of 3 evidence-based, CBT-framed exercises: received support & cognitive distortions, social skills & peer support, and action planning. Participants will have an option to engage in one or more out of four additional modules: relaxation, cognitive reconstruction, mindfulness, and lifestyle. The condition takes 3 weeks, 1 week per exercise.
  Arms: Perceived Social Support

SUMMARY:
The aim of this study is to assess the efficacy of internet intervention for reduction of occupational stress and its negative consequences (job burnout, depression) among medical professionals through the enhancement of the resources that are critical for coping with stress: self-efficacy and perceived social support.

DETAILED DESCRIPTION:
Medical professionals are at high risk for job stress and burnout. Research show that the negative effects of stress can be reduced through strengthening personal resources such as self-efficacy and perceived social support. In line with cultivation and enabling hypotheses (Schwarzer & Knoll, 2007; Benight & Bandura, 2004) either self-efficacy cultivates perceived support, or rather perceived support enables self-efficacy. This study aims at testing both hypotheses in experimental design by applying them as a theoretical framework for the Med-Stress: evidence-based, CBT-framed internet intervention to foster resource accumulation among medical professionals.

The effectiveness of intervention will be tested in a four-arm randomized controlled trial comparing the effects of: 1) self-efficacy and perceived support sequential enhancement (cultivation hypothesis), 2) perceived support and self-efficacy sequential enhancement (enabling hypothesis), 3) only self-efficacy, and 4) only social support enhancement (controls). Primary outcomes are job stress and burnout, secondary outcomes include work engagement, depression, and secondary traumatic stress. Self-efficacy and perceived support are expected to mediate the relationships between condition assignment and outcomes. Assessments include baseline (T1), three- or six-weeks post-test (depending on the condition, T2), as well as six- and twelve-months follow-ups (T3, T4). Intervention effect sizes and between-groups comparisons at post-test and follow-ups will be calculated.

This study will contribute to the findings on the role of personal resources in the development of job stress and burnout by demonstrating the cultivation vs enabling effects of self-efficacy and perceived social support.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Professionally active medical providers
* Internet connection

Exclusion Criteria:

* No access to a device with Internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change on Perceived Stress Scale 14 (PSS-14) | Change from baseline on PSS-14 (3 or 6 weeks depending on the study condition)
  The PSS-14 is a measure of perceived stress. It consists of 14 items with response scale ranging from 0 to 4. Higher total score represents higher perceived stress. Instruction was adapted to refer to work-related stress.
Change on Perceived Stress Scale 14 (PSS-14) | Change from baseline on PSS-14 (6 months)
  The PSS-14 is a measure of perceived stress. It consists of 14 items with response scale ranging from 0 to 4. Higher total score represents higher perceived stress. Instruction was adapted to refer to work-related stress.
Change on Perceived Stress Scale 14 (PSS-14) | Change from baseline on PSS-14 (12 months)
  The PSS-14 is a measure of perceived stress. It consists of 14 items with response scale ranging from 0 to 4. Higher total score represents higher perceived stress. Instruction was adapted to refer to work-related stress.
Change on Oldenburg Burnout Inventory (OLBI) | Change from baseline on OLBI (3 or 6 weeks depending on the study condition)
  The OLBI is a measure of job burnout. It consists of 16 items with response scale ranging from 1 to 4. The questionnaire consists of two subscales: exhaustion and disengagement, To compute total score subscales are summed. Higher total score represents higher job burnout.
Change on Oldenburg Burnout Inventory (OLBI) | Change from baseline on OLBI (6 months)
  The OLBI is a measure of job burnout. It consists of 16 items with response scale ranging from 1 to 4. The questionnaire consists of two subscales: exhaustion and disengagement, To compute total score subscales are summed. Higher total score represents higher job burnout.
Change on Oldenburg Burnout Inventory (OLBI) | Change from baseline on OLBI (12 months)
  The OLBI is a measure of job burnout. It consists of 16 items with response scale ranging from 1 to 4. The questionnaire consists of two subscales: exhaustion and disengagement, To compute total score subscales are summed. Higher total score represents higher job burnout.

SECONDARY OUTCOMES:
Change on Utrecht Work Engagement Scale (UWES-3) | Change from baseline on UWES-3 (3 or 6 weeks depending on the study condition)
  The UWES-3 is a measure of work engagement. It consists of 3 items with response scale ranging from 0 to 6. Higher total score represents higher work engagement.
Change on Utrecht Work Engagement Scale (UWES-3) | Change from baseline on UWES-3 (6 months)
  The UWES-3 is a measure of work engagement. It consists of 3 items with response scale ranging from 0 to 6. Higher total score represents higher work engagement.
Change on Utrecht Work Engagement Scale (UWES-3) | Change from baseline on UWES-3 (12 months)
  The UWES-3 is a measure of work engagement. It consists of 3 items with response scale ranging from 0 to 6. Higher total score represents higher work engagement.
Change on Patient Health Questionnaire (PHQ-9) | Change from baseline on PHQ-9 (3 or 6 weeks depending on the study condition)
  The PHQ-9 is a measure of depression. It consists of 9 items with response scale ranging from 0 to 3. Higher total score represents higher depression.
Change on Patient Health Questionnaire (PHQ-9) | Change from baseline on PHQ-9 (6 months)
  The PHQ-9 is a measure of depression. It consists of 9 items with response scale ranging from 0 to 3. Higher total score represents higher depression.
Change on Patient Health Questionnaire (PHQ-9) | Change from baseline on PHQ-9 (12 months)
  The PHQ-9 is a measure of depression. It consists of 9 items with response scale ranging from 0 to 3. Higher total score represents higher depression.
Change on Posttraumatic Stress Disorder Checklist 5 (PCL-5) | Change from baseline on PCL-5 (3 or 6 weeks depending on the study condition)
  The PCL-5 is a measure of posttraumatic stress disorder. It consists of 20 items with response scale ranging from 0 to 4. The questionnaire consists of four subscales: intrusions, avoidance, negative alterations in cognition and mood, and arousal. To compute total score subscales are summed. Higher total score represents higher posttraumatic stress disorder. Instruction was adapted to refer to work-related secondary traumatic stress.
Change on Posttraumatic Stress Disorder Checklist 5 (PCL-5) | Change from baseline on PCL-5 (6 months)
  The PCL-5 is a measure of posttraumatic stress disorder. It consists of 20 items with response scale ranging from 0 to 4. The questionnaire consists of four subscales: intrusions, avoidance, negative alterations in cognition and mood, and arousal. To compute total score subscales are summed. Higher total score represents higher posttraumatic stress disorder. Instruction was adapted to refer to work-related secondary traumatic stress.
Change on Posttraumatic Stress Disorder Checklist 5 (PCL-5) | Change from baseline on PCL-5 (12 months)
  The PCL-5 is a measure of posttraumatic stress disorder. It consists of 20 items with response scale ranging from 0 to 4. The questionnaire consists of four subscales: intrusions, avoidance, negative alterations in cognition and mood, and arousal. To compute total score subscales are summed. Higher total score represents higher posttraumatic stress disorder. Instruction was adapted to refer to work-related secondary traumatic stress.

OTHER OUTCOMES:
Change on Work Stress and Job Burnout Self-Efficacy Scale (WSBSES) | Change from baseline on WSBSES (3 or 6 weeks depending on the study condition)
  The WSBSES is a measure of self-efficacy to cope with work stress and job burnout. It consists of 28 items with the response scale ranging from 1 to 7. Higher total score represents higher self-efficacy.
Change on Work Stress and Job Burnout Self-Efficacy Scale (WSBSES) | Change from baseline on WSBSES (6 months)
  The WSBSES is a measure of self-efficacy to cope with work stress and job burnout. It consists of 28 items with the response scale ranging from 1 to 7. Higher total score represents higher self-efficacy.
Change on Work Stress and Job Burnout Self-Efficacy Scale (WSBSES) | Change from baseline on WSBSES (12 months)
  The WSBSES is a measure of self-efficacy to cope with work stress and job burnout. It consists of 28 items with the response scale ranging from 1 to 7. Higher total score represents higher self-efficacy.
Change on Berlin Social Support Scales (BSSS), Subscale 3 | Change from baseline on BSSS, Subscale 3 (3 or 6 weeks depending on the study condition)
  The BSSS Subscale 3 measures social support seeking. Instruction and rating scale ware adapted to refer to social support self-efficacy. It consists of 5 items with response scale ranging from 1 to 7. Higher total score represents higher social support self-efficacy.
Change on Berlin Social Support Scales (BSSS), Subscale 3 | Change from baseline on BSSS, Subscale 3 (6 months)
  The BSSS Subscale 3 measures social support seeking. Instruction and rating scale ware adapted to refer to social support self-efficacy. It consists of 5 items with response scale ranging from 1 to 7. Higher total score represents higher social support self-efficacy.
Change on Berlin Social Support Scales (BSSS), Subscale 3 | Change from baseline on BSSS, Subscale 3 (12 months)
  The BSSS Subscale 3 measures social support seeking. Instruction and rating scale ware adapted to refer to social support self-efficacy. It consists of 5 items with response scale ranging from 1 to 7. Higher total score represents higher social support self-efficacy.
Change on Who Can You Count On Scale | Change from baseline on Who Can You Count On Scale (3 or 6 weeks depending on the study condition)
  The scale measures perceived social support. It consists of 32 items with response scale ranging from 1 to 5. The questionnaire consists of 4 subscales: support form supervisors, support from friends, support from family, friends. To compute total score subscales are summed. Higher total score represents higher perceived social support.
Change on Who Can You Count On Scale | Change from baseline on Who Can You Count On Scale (6 months)
  The scale measures perceived social support. It consists of 32 items with response scale ranging from 1 to 5. The questionnaire consists of 4 subscales: support form supervisors, support from friends, support from family, friends. To compute total score subscales are summed. Higher total score represents higher perceived social support.
Change on Who Can You Count On Scale | Change from baseline on Who Can You Count On Scale (12 months)
  The scale measures perceived social support. It consists of 32 items with response scale ranging from 1 to 5. The questionnaire consists of 4 subscales: support form supervisors, support from friends, support from family, friends. To compute total score subscales are summed. Higher total score represents higher perceived social support.
Secondary Trauma Exposure Scale (STES) | Baseline
  The STES measures job-related indirect exposure to traumatic events. It consists of 12 items with response scale for 10 items ranging from 0 to 1 and for remaining 2 items from 0 to 7. Higher total score represents higher secondary trauma exposure.
Credibility and Expectancy Questionnaire (CEQ) | Baseline
  The CEQ measures expectancy and credibility of the intervention. It consists of 6 items, with response scale for 4 items ranging from 1 to 9, and for remaining 2 items from 0% to 100%. Higher total score represents higher treatment credibility and user's expectancy for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ewelina Smoktunowicz, PhD, Principal Investigator — SWSP University of Social Sciences and Humanities, Department of Psychology
Locations (1):
- SWPS University of Social Sciences and Humanities, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benight CC, Bandura A. Social cognitive theory of posttraumatic recovery: the role of perceived self-efficacy. Behav Res Ther. 2004 Oct;42(10):1129-48. doi: 10.1016/j.brat.2003.08.008. PMID 15350854
- [Background] Cieslak R, Anderson V, Bock J, Moore BA, Peterson AL, Benight CC. Secondary traumatic stress among mental health providers working with the military: prevalence and its work- and exposure-related correlates. J Nerv Ment Dis. 2013 Nov;201(11):917-25. doi: 10.1097/NMD.0000000000000034. PMID 24177477
- [Background] Widerszal-Bazyl M, Cieslak R. Monitoring psychosocial stress at work: development of the Psychosocial Working Conditions Questionnaire. Int J Occup Saf Ergon. 2000;Spec No:59-70. doi: 10.1080/10803548.2000.11105108. PMID 10828153
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Demerouti E, Mostert K, Bakker AB. Burnout and work engagement: a thorough investigation of the independency of both constructs. J Occup Health Psychol. 2010 Jul;15(3):209-222. doi: 10.1037/a0019408. PMID 20604629
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lua H.J. The mediating role of work stress and burnout management self-efficacy in the job demand - resources model [dissertation]. SWPS University of Social Sciences and Humanities, Warsaw 2008.
- [Background] Schaufeli, W.B., Shimazu, A., Hakanen, J., Salanova, M., & De Witte, H. (2017). An ultra-short measure for work engagement: The UWES-3. Validation across five countries. European Journal of Psychological Assessment. Advance online publication. doi:10.1027/1015-5759/a000430.
- [Background] Schwarzer, R., & Knoll, N. (2007). Functional roles of social support within the stress and coping process: A theoretical and empirical overview. International journal of psychology, 42(4), 243-252. doi: 10.1080/00207590701396641
- [Background] Schwarzer R, Schulz U (2000) Berlin Social Support Scale (BSSS). Retrieved from http://userpage.fu-berlin.de/~health/bsss.htm
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Derived] Smoktunowicz E, Lesnierowska M, Carlbring P, Andersson G, Cieslak R. Resource-Based Internet Intervention (Med-Stress) to Improve Well-Being Among Medical Professionals: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 11;23(1):e21445. doi: 10.2196/21445. PMID 33427674
- [Derived] Smoktunowicz E, Lesnierowska M, Cieslak R, Carlbring P, Andersson G. Efficacy of an Internet-based intervention for job stress and burnout among medical professionals: study protocol for a randomized controlled trial. Trials. 2019 Jun 10;20(1):338. doi: 10.1186/s13063-019-3401-9. PMID 31182128